CLINICAL TRIAL: NCT02718313
Title: Echocardiographic Findings and 30-days Outcomes for Intraventricular Conduction Delay in Patients Undergoing Elective Surgeries
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0005
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: General Anesthesia
Keywords: intraventricular conduction delay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intraventricular conduction delay: Transthoracic echocardiography will be performed to investigate whether the patients have the cardiac disease or not. The transthoracic echocardiography will be performed after the induction of general anesthesia and before the start of surgery.

SUMMARY:
The purpose of this study is to investigate the type of the cardiac disease using transthoracic echocardiography in patients whose preoperative electrocardiography shows the intraventricular conduction delay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged over 20 yrs who are scheduled for surgery under the general anesthesia and whose preoperative electrocardiography finding is intraventricular conduction delay.

Exclusion Criteria:

* Patients who are planning cardiac surgery
* Patients who has chest wall disease
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients who are planning surgery under general anesthesia and whose preoperative electrocardiography reading is intraventricular conduction delay
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
presence of cardiac disease | Within 1 hour after the induction of general anesthesia
  Transthoracic echocardiography will be performed to investigate the evidence of the cardiac disease after the induction of general anesthesia and before the start of the surgery.

IPD SHARING:
Plan to Share IPD: No
no plan to share data